CLINICAL TRIAL: NCT03998787
Title: Metabotropic Receptors For Glutamate Type 3 In Parkinson's Disease: Clinical And Neurophysiological Correlations
Brief Title: Metabotropic Receptors For Glutamate Type 3 In Parkinson's
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Alfredo Berardelli, Pincipal Investigator, Neuromed IRCCS
Other Study IDs: ALBE_01
Record Dates: First submitted 2019-06-14; First posted 2019-06-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Neuroscience; Movement Disorders
Keywords: Parkinson's disease; Neurophysiology
MeSH Terms: conditions — Movement Disorders; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Parkinson's disease: Patients with Parkinson's disease
  Interventions: Other: Neurophysiological assessment
- Healthy Subjects: Healthy subjects
  Interventions: Other: Neurophysiological assessment

INTERVENTIONS:
Other: Neurophysiological assessment — Kinematic analysis of movement and transcranial magnetic stimulation

SUMMARY:
Parkinson's disease (PD) is characterized by bradykinesia, rigidity, and tremor. Several scientific pieces of evidence, based on the use of kinematic techniques, have allowed quantifying objectively the alterations of the voluntary movement in the different stages of the disease. In recent years, several studies using transcranial magnetic stimulation (TMS) techniques, have also shown abnormalities in neurophysiological parameters of the primary motor cortex (M1) in patients with MP, in particular, a reduction in cortical excitability and synaptic plasticity of M1. In addition to the central role played by a dopaminergic deficit in MP, recent evidence suggests a possible involvement of the neurotransmitter glutamatergic system. In the present monocentric observational study, the investigators propose to assess possible correlations between polymorphisms of metabotropic glutamate type 3 receptors (mGlu3), clinical evaluation scales, alterations of kinematic motion parameters and neurophysiological parameters of M1.

DETAILED DESCRIPTION:
In recent years, numerous neurophysiological studies have characterized the alterations of voluntary movement and the pathophysiological mechanisms of MP. Kinematic studies have shown that in addition to bradykinesia, which literally means slowing of movement, voluntary movements in PD are characterized by reduced amplitude (hypokinesia), altered rhythmicity (dysrhythmia) and progressive decrease in amplitude and speed during the execution of repetitive movements (sequence effect). Recent evidence also suggests that the characteristics of voluntary movement can vary in the various stages of PD, it has been observed, for example, that in early stages of disease, i.e. in newly diagnosed patients not previously treated with dopaminergic drugs repetitive finger-tapping movements are characterized by reduced amplitude and speed and the effect sequence, without significant changes in the rhythm of movement. In the advanced stages of PD, movement is characterized by a marked decrease in amplitude and velocity and by an altered rhythm of movement but not by the sequence effect.

TMS is a neurophysiological technique that allows the non-invasive study of different physiological mechanisms of M1 in humans. Stimulation, delivered in single stimuli, allows for example to evaluate neurophysiological parameters such as motor thresholds, the amplitude of motor evoked potentials (MEPs) and the so-called input-output recruitment curve of MEPs, i.e. parameters that reflect the overall excitability of the corticospinal system. TMS delivered in pairs of magnetic stimuli allows additional parameters to be evaluated, such as intracortical inhibition at short intervals (SICI) and intracortical facilitation (ICF), i.e. parameters that reflect the excitability of inhibitory and facilitator cortical interneurons. In recent years, further protocols have been developed using the repetitive stimulation of M1 to induce lasting changes in the amplitude of MEPs that are thought to reflect the mechanisms of synaptic plasticity, similar to similar phenomena observed in the experimental animal. In particular, the technique of associative stimulation (PAS), is based on percutaneous electrical stimulation of the peripheral nerve and concomitant stimulation of M1 by TMS at certain inter-stimulation intervals (25ms or 10ms) to induce lasting changes, in a facilitatory or inhibitory sense, in the amplitude of MEPs. Numerous TMS studies have been performed in PD patients in recent years. Among the main results observed are altered excitability of M1, especially a reduced SICI and reduced synaptic plasticity, tested with the PAS technique or other methods. Recently, we have also observed that some alterations of excitability and plasticity of M1 correlate with specific kinematic alterations of movement in PD patients, suggesting therefore that neurophysiological changes of M1 contribute to the pathophysiology of bradykinesia. In addition to the central role played by a dopaminergic deficit in MP, recent evidence suggests a possible involvement of the neurotransmitter glutamatergic system.

MAIN ASSUMPTIONS AND OBJECTIVES

Hypothesis:

Previous studies have observed relationships between the reduced cortical inhibition and reduced synaptic plasticity of M1 and the overall severity of PD evaluated with standardized clinical scales and kinematic motion analysis techniques. In the present study, we will relate metabotropic type 3 glutamate receptor polymorphisms (mGlu3) to the severity of motor and non-motor symptoms, cortical plasticity and other neurophysiological parameters in patients with PD.

Preliminary data:

Previous observations obtained in our laboratory have shown that the kinematic study in PD is a valid technique for objectively documenting various alterations of voluntary movement, including bradykinesia, hypokinesia, altered rhythmicity, and sequence effect. These characteristics may change at various stages of PD. For example, it has been observed that in the early stages of illness, repetitive finger movements are characterized by reduced amplitude and speed and by the sequence effect, without significant alterations in the rhythm of the movement. In the advanced stages of PD, movement is characterized by a marked decrease in amplitude and velocity and an altered rhythm of movement but not by the sequence effect. Kinematic studies in patients with PD have also made it possible to objectively quantify the effects of dopaminergic replacement therapy on the various alterations that characterize the PD. The objective effects of dopaminergic therapy on the various alterations of voluntary movement, quantified by kinematic studies, are variable. In particular, it has been repeatedly observed that the sequencing effect in patients with PD does not improve significantly following the administration of dopaminergic drugs. Previous observations obtained in TMS studies have also demonstrated altered M1 excitability in patients with PD, including for example reduced SICI and reduced synaptic plasticity, tested with the PAS technique or other methods. In some cases, it has been observed that the administration of dopaminergic drugs is able to normalize the alterations of neurophysiological parameters of M1 in PD, the results are however variable. Recently, we have observed that some alterations of excitability and plasticity of M1 correlate with specific kinematic alterations of movement in PD patients, suggesting therefore that neurophysiological changes of M1 contribute to the pathophysiology of bradykinesia.

Objectives:

In the present monocentric observational study, the investigators propose to:

A) To carry out an accurate characterization of the alterations of the voluntary movement in patients with PD through the use of standardized clinical scales and a computerized system for the objective analysis of the voluntary movement and a detailed study of possible neurophysiological alterations of M1 in patients with PD, through the use of TMS techniques.

B) Evaluate metabotropic type 3 glutamate receptor polymorphisms (mGlu3) in PD patients.

C) Investigate possible correlations between type 3 metabotropic glutamate receptor polymorphisms (mGlu3), clinical evaluation scales, alterations of kinematic motion parameters and neurophysiological parameters of M1.

METHODOLOGY AND EXPERIMENTAL DESIGN The study involves the recruitment of 20 PD patients, diagnosed according to current clinical criteria and 20 healthy control subjects. Patients with motor fluctuations and dyskinesia will be excluded. Recruitment of patients and control subjects will be carried out at the IRCCS NEUROMED Institute, Pozzilli (IS). All PD patients will undergo blood sampling to assess metabotropic glutamate type 3 (mGlu3) receptor polymorphisms All study participants will give informed consent to the experimental procedures, which will be approved by the local ethics committee and conducted in accordance with the Helsinki Declaration.

Standardized clinical scales and a computerized system for objective analysis of voluntary movement will be used to characterize alterations of voluntary movement in PD patients. With this system, the movements of the upper limb will be examined, following the instructions dictated by the scale most widely used today in the clinical environment, namely the new version of the UPDRS, promoted by the Movement Disorder Society. The repetitive movements of the fingers will be examined by inviting the patient to tap his index finger on his thumb. For each test, the movements shall be made for 15 seconds in succession. Three recordings will be made for each movement. Participants will be encouraged to make the movements as fast and as wide as possible. The movements will be analyzed at the most affected side. The computerized analysis system will allow to objectively extrapolate the parameters related to speed, amplitude, the rhythm of the movement and effect-sequence.

The study of neurophysiological alterations of M1 will be carried out by means of the TMS technique. Ejecting single magnetic stimuli, a measurement of parameters reflecting the excitability of the corticospinal pathway will be carried out, i.e. the measurement of motor thresholds and of the input-output recruitment curve. By delivering magnetic stimuli in pairs, according to a condition-test paradigm, at inter-stimulus intervals fixed at 2-4-10 and 15ms parameters reflecting the excitability of intracortical circuits of inhibitory (SICI) and facilitatory (ICF) type will be measured. Finally, the PAS technique will be used to study the mechanisms of synaptic plasticity of M1. PAS uses joint peripheral nerve stimulation (percutaneous electrical stimulation) and M1 (TMS) at an inter-stimulation interval fixed at 25ms. During the PAS technique, 225 stimuli are delivered globally, at a frequency of 0.4 Hz and for a total duration of 15 minutes of stimulation.

Patients with PD will be studied in a single experimental session, at least twelve hours after the suspension of dopaminergic drugs (OFF session). Healthy control subjects will be evaluated in a single experimental session.

MEANING AND INNOVATION The main innovative aspect of the study is the integrated approach that involves the use of both techniques of kinematic analysis of movement, and techniques of non-invasive brain stimulation. The present work could, therefore, allow to deepen the current knowledge and to obtain advancement in terms of understanding the pathophysiological mechanisms underlying the altered motor control in patients with PD.

EQUIPMENT AND RESOURCES The study will be carried out at the IRCCS NEUROMED Institute, Pozzilli (IS). The institute has the material to conduct the study and in particular: the optoelectronic system of infrared cameras (sampling rate, 120Hz), (SMART motion system, BTS Engineering, Milan, Italy) for kinematic evaluation; the dedicated software for kinematic data analysis (SMART Analyzer, BTS Engineering, Milan, ltaly); two Magstim magnetic stimulators (Magstim Company, Withland, UK) for single and double stimulation magnetic stimulation and one DS7 Digitimer electric simulator (Digitimer, UK) for PAS stimulation; one D 360 Digitimer amplifier (Digitimer, UK) and one AD 1401 plus analogue-to-digital converter (Cambridge Electronic Design, UK) for recording the electromyographic signal; one dedicated software (Signal® version 4.00, Cambridge Electronic Design, UK) for off-line analysis of the electromyographic signal.

TRANSLATIONAL RELEVANCE OF THE STUDY The results of the study could be useful for a better understanding of the pathophysiological mechanisms, and in particular of the involvement of M1, at the basis of the alterations of voluntary movement in MP. The results of the study could also be useful in developing possible treatments, based on the use of subtype-selective agonists and positive allosteric modulators of metabotropic glutamate type 3 receptors (mGlu3).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Must be able to participate to the experimental session

Exclusion Criteria:

* Controindications to transcranial magnetic stimulation.
* Presence of dyskinesias

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study involves the recruitment of 20 patients with Parkinson's disease, diagnosed according to current clinical criteria and 20 healthy control subjects. Patients with motor fluctuations and dyskinesia will be excluded. Recruitment of patients and control subjects will be carried out at the IRCCS NEUROMED Institute, Pozzilli (IS). All patients will undergo blood sampling to assess polymorphisms of metabotropic glutamate type 3 (mGlu3) receptors. All study participants will give informed consent to the experimental procedures, which will be approved by the local ethics committee and conducted in accordance with the Helsinki Declaration.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological assessment of PD patients | 1 hours
  Kinematic analysis of movement (i.e. amplitude and velocity)
Neurophysiological assessment of PD patients | 1 hour
  Transcranial magnetic stimulation of primary motor cortex (i.e. aamplitude of motor evoked potentials)

SECONDARY OUTCOMES:
Genetic analysis | 5 minutes
  Metabotropic glutamate type 3 receptor polymorphisms analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berardelli, Principal Investigator — IRCCS Neuromed

IPD SHARING:
Plan to Share IPD: Undecided